CLINICAL TRIAL: NCT02664207
Title: Extended Criteria For Fetal Myelomeningocele Repair: A Pilot Study
Brief Title: Extended Criteria For Fetal Myelomeningocele Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, KuoJen Tsao, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-15-0795
Record Dates: First submitted 2016-01-19; First posted 2016-01-26 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Obesity; Myelomeningocele; Pregnancy; Diabetes Mellitus in Pregnancy; Fetal Anomaly
Keywords: Myelomeningocele repair; Open Neural Tube Defect; BMI of 35-40 kg/m2,; Open Fetal Surgery; Elevated body mass index
MeSH Terms: conditions — Obesity; Meningomyelocele; Diabetes, Gestational; Congenital Abnormalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fetal Surgery in Women with ex (Experimental): Fetal myelomeningocele repair surgery will be offered to pregnant women meeting the criteria for surgery (as set by the MOMS trial) with the exception of the following:
  * a BMI greater than 35 (but less than or equal to 40 kg/m2)
  * (minor) Fetal structural abnormality
  * (well-controlled) Diabetes
  * Previous preterm delivery (followed by a full term delivery)
  * Maternal red cell alloimmunization (must NOT be associated with fetal disease, OR fetus must have negative red cell antigen status as determined by amniocentesis).
  Intervention: Open Fetal Repair of Myelomeningocele
  Interventions: Procedure: Open Fetal Repair of Myelomeningocele

INTERVENTIONS:
Procedure: Open Fetal Repair of Myelomeningocele — Fetal repair of myelomeningocele in women with additional medical factors that would have excluded them from this treatment under the MOMs trial inclusion/exclusion criteria

SUMMARY:
The purpose of this study is to offer pre-natal Myelomeningocele (MMC) repair surgery to pregnant women with one of the former surgery exclusion factors

* A BMI of 35-40 kg/m2
* Diabetes; patients will require good glycemic control
* History a previous preterm birth, as long as it was followed by a full term birth
* Structural abnormality in the fetus; abnormality must be minor, not increasing the risk of prematurity. For example cleft lip and palate, minor ventricular septal defect, pyelectasis.
* Maternal Rh alloimmunization. Must have a low level of anti-red blood cell antibody that is not associated with fetal disease, specifically anti-E < 1:4 or anti-M. Or alloimmunization with negative fetal red blood cell antigen status determined by amniocentesis.

We will be extending the Management of Myelomeningocele Study (MOMs) criteria by including these factors. Prenatal clinical and outcome information will be collected; safety and efficacy will be evaluated

DETAILED DESCRIPTION:
The purpose of this study is to extend the MOMs requirements for pre-natal MMC repair surgery and evaluate safety and efficacy. This will be accomplished through prenatal and post-operative observation and data collection.

The data collected will be documented and collected from prenatal ultrasounds, operative, and delivery reports. We will share our preliminary data with NAFTNet in order to prompt a multicenter trial; this collaboration will help propagate further research and answer clinical questions regarding this extension in surgery criteria.

ELIGIBILITY:
Inclusion Criteria:

* Any woman with a prenatal diagnoses of myelomeningocele.
* Pre-pregnancy BMI of 35-45 kg/m2.
* Diabetes; patients will require good glycemic control
* History a previous preterm birth, as long as it was followed by a full term birth
* Structural abnormality in the fetus; abnormality must be minor, not increasing the risk of prematurity. For example cleft lip and palate, minor ventricular septal defect, pyelectasis.
* Maternal Rh alloimmunization. Must have a low level of anti-red blood cell antibody that is not associated with fetal disease, specifically anti-E < 1:4 or anti-M. Or alloimmunization with negative fetal red blood cell antigen status determined by amniocentesis.
* same MOMs Trial inclusion criteria with the exception of the above.

Exclusion Criteria:

* poor glycemic control (i.e., HbA1c ≥ 8%) in spite a medical antidiabetic therapy in accordance with good clinical practice (GCP)
* presence of significant co-morbidities or complications (such as dyslipidemia, uncontrolled arterial hypertension, impaired renal function, neuropathy, retinopathy, CVD)
* severe diabetes complications or associated medical conditions (such as blindness, endstage renal failure, liver cirrhosis, malignancy, chronic congestive heart failure)
* recent (within preceding 12 months) myocardial infarction, stroke or TIA
* unstable angina pectoris
* same MOMs Trial exclusion criteria (with the exception of extended inclusion criteria)

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2016-01-26; Primary Completion 2023-12 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Post-operative complications | At the time of fetal repair surgery to 40 weeks gestation
  Determine if there is an increased risk in women in this group

CONTACTS AND LOCATIONS:
Overall Officials: Kuojen Tsao, MD, Principal Investigator — The University of Texas Health Science Center at Houston - UTHealth.
Locations (2):
- United States (2):
  - Children's Memorial Hermann Hospital, Houston, Texas
  - The Fetal Center at UTHealth, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Adzick NS, Thom EA, Spong CY, Brock JW 3rd, Burrows PK, Johnson MP, Howell LJ, Farrell JA, Dabrowiak ME, Sutton LN, Gupta N, Tulipan NB, D'Alton ME, Farmer DL; MOMS Investigators. A randomized trial of prenatal versus postnatal repair of myelomeningocele. N Engl J Med. 2011 Mar 17;364(11):993-1004. doi: 10.1056/NEJMoa1014379. Epub 2011 Feb 9. PMID 21306277
- See also: The Fetal Center at Children's Memorial Hermann Hospital — http://childrens.memorialhermann.org/the-fetal-center/